CLINICAL TRIAL: NCT06375161
Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Infusion of Anti-CD19-CAR-T Cells in Relapsed/Refractory B-cell Tumor Patients.
Brief Title: Anti-CD19-CAR-T Cells in Relapsed/Refractory B-cell Tumor Patients.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., professor,Chief Physician,Vice President of Tongji Hospital, Tongji University School of Medicine etc., Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CN-A6
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-08

CONDITIONS: B Cell Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19-CAR-T Cells (Experimental): anti-CD19-CAR-T cell infusion. Infusion doses: The planned infusion doses are as follows: the first dose group at 1×10^5 cells/kg; the second dose group at 3×10^5 cells/kg; the third dose group at 1×10^6 cells/kg. Infusion doses refer to the number of CAR-positive cells.
  Administration route: anti-CD19-CAR-T cells are administered via intravenous drip at a rate of approximately 2 to 5 mL/minute using an infusion pump, with a recommended infusion time of less than 30 minutes.
  Interventions: Biological: anti-CD19-CAR-T cells

INTERVENTIONS:
Biological: anti-CD19-CAR-T cells — Before cell infusion, Investigator may decide, based on necessity, whether to administer prophylactic medication, which may include options such as acetaminophen and diphenhydramine, or H1 antihistamines, among others.
  Subjects are allowed to receive adequate supportive care after anti-CD19-CAR-T cell infusion, including blood transfusions and blood products, antibiotic therapy, antiemetics, antidiarrheals, analgesics, etc.

SUMMARY:
This study is a single-center, open-label, single-dose clinical trial of anti-CD19-CAR-T cell therapy in relapsed/refractory B-cell tumor patients after Qinglin pre-treatment.

In this study phase, a traditional "3+3" trial design is employed for dose escalation.

DETAILED DESCRIPTION:
The study plans to include CD19-positive relapsed/refractory B-cell tumor patients. After the screening period, peripheral blood mononuclear cell (PBMC) collection, and lymphocyte depletion pre-treatment period, subjects will receive a single infusion of anti-CD19-CAR-T cells. In addition to the baseline period, efficacy assessments will be conducted monthly for ALL subjects and at weeks 4, 12, 24, 36, and 48 post-treatment for NHL subjects, until disease progression (PD), relapse, change of treatment regimen, death, intolerable toxicity, at the discretion of the investigator, or voluntary withdrawal by the patient (whichever occurs first).

Toxicity will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Safety of anti-CD19-CAR-T cell therapy will be evaluated through laboratory tests, 12-lead electrocardiograms, vital signs, physical examinations, etc. Blood samples will be collected from subjects to assess cellular pharmacokinetics and explore the effects of cellular drugs on ferritin, C-reactive protein, and related cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical trial; the individual or legal guardian fully understands and consents to the study by signing the Informed Consent Form (ICF); willing and able to comply with all trial procedures.
2. Age between 18-70 years.
3. Patients who are refractory or relapsed after current standard treatments (including allogeneic or autologous hematopoietic stem cell transplantation), and not suitable for other treatment options such as a second hematopoietic stem cell transplantation.

   1. Relapsed/refractory B-cell acute lymphoblastic leukemia (ALL) is defined as one of the following:

      - Primary refractory disease

      - First relapse if the first remission was ≤12 months
      * Relapse or refractory disease after two or more lines of systemic therapy
      * Relapse or refractory disease after allogeneic transplantation, provided that at least 100 days have elapsed since transplantation at the time of enrollment, and no immunosuppressive drugs have been used for at least 4 weeks prior to enrollment, except for low-dose steroids (≤5 mg prednisone or equivalent).
   2. Subjects with Ph+ B-cell ALL who are intolerant or ineligible for treatment with tyrosine kinase inhibitors (TKIs), or have relapsed/refractory disease after receiving at least two different TKI treatments, are eligible.
   3. Relapsed/refractory B-cell non-Hodgkin lymphoma (NHL) is defined as one of the following:

      1. No response to first-line treatment (primary refractory disease); excluding subjects intolerant to first-line chemotherapy - PD as the best response to first-line treatment - Best response after at least 4 cycles of first-line treatment (such as 4 cycles of RCHOP) is SD, and the duration of SD after the last dose does not exceed 6 months.
      2. No response to second-line or subsequent treatments - PD as the best response to the most recent treatment regimen - Best response after at least 2 cycles of last-line treatment is SD, and the duration of SD after the last dose does not exceed 6 months.
      3. Refractory after ASCT

         - Disease progression or relapse ≤12 months post-ASCT (relapse must be confirmed by biopsy).
         * If salvage therapy is given post-ASCT, subjects must have had no response or relapse after the last-line treatment.
4. Bone marrow smear reports showing tumor cells ≥5% in ALL patients.
5. Patients with refractory or relapsed NHL meet one of the following subtypes:

1) DLBCL-NOS. 2) Primary mediastinal large B-cell lymphoma (PMBCL). 3) Transformed follicular lymphoma (TFL), previously treated with follicular lymphoma chemotherapy, subsequently transformed into refractory disease after DLBCL.

4) Mantle cell lymphoma. 5) High-grade B-cell lymphoma. 6) CLL/SLL.

(6) ECOG performance status ≤2.

(7) Estimated life expectancy of at least 12 weeks.

(8) Adequate venous access (for single collection) and no other contraindications to blood cell separation.

(9) Laboratory test results at screening must meet the following requirements, and subjects must not have received colony-stimulating factors (G-CSF/PEG-CSF) within 2 weeks prior to hematological assessment (except for low-dose steroids):

1) Absolute neutrophil count ≥1.0×10^9/L, ALL eligibility to be determined by the investigator.

2) Hemoglobin ≥60 g/L (without red blood cell transfusion within 14 days). 3) Platelets ≥50×10^9/L, ALL eligibility to be determined by the investigator. 4) Absolute lymphocyte count (ALC) ≥ 0.5×10^9/L; if insufficient, and T-cell proportion is high in the lymphocyte subset, the investigator can discuss with the sponsor.

5) Serum total bilirubin ≤1.5× upper limit of normal (ULN). 6) Aspartate transaminase (AST), alanine transaminase (ALT) ≤2.5× ULN. 7) Creatinine <1.5× ULN and creatinine clearance ≥60 mL/minute.

(10) Left ventricular ejection fraction ≥45%, echocardiography (ECHO) confirms no clinically significant pericardial effusion (except for trace or physiological), and electrocardiography results have no clinical significance.

(11) Baseline oxygen saturation in room air >92%.

(12) Women of childbearing potential must have negative serum or urine pregnancy tests (women who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered women of childbearing potential).

Exclusion Criteria:

(1) ALL with central nervous system abnormalities, excluding clinically evident neurological changes CNS-2 and CNS-3.

1) CNS-3 disease, defined as detectable tumor cells in the cerebrospinal fluid (CSF), with ≥5 WBCs per mm3, with or without neurological changes.

2) CNS-2 disease, defined as detectable tumor cells in the CSF, with <5 WBCs per mm3, and neurological changes.

Note: Subjects with CNS-1 (no tumor cells detected in CSF) and CNS-2 with no clinically evident neurological changes are eligible for this study.

(2) Evidence of central nervous system lymphoma on brain MRI; active primary central nervous system DLBCL, unless the central nervous system involvement has been effectively treated (i.e., participants are asymptomatic), and >4 weeks have elapsed since local treatment before enrollment.

(3) Active central nervous system diseases such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any autoimmune diseases involving the central nervous system.

(4) History of or concurrent malignancies other than CD19+ malignancies.

(5) Clinically significant cardiac diseases, or arrhythmias not controlled by medication.

(6) Presence or suspicion of uncontrolled fungal, bacterial, viral, or other infections, or requiring intravenous antibiotic therapy; simple urinary tract infections and uncomplicated bacterial pharyngitis are allowed if responsive to treatment and after consultation with the sponsor's medical monitor.

(7) Hepatitis B (positive for hepatitis B surface antigen and/or positive for hepatitis B core antibody with hepatitis B DNA >1000 copies/ml) and hepatitis C (positive for hepatitis C antibody); syphilis, human immunodeficiency virus (HIV) infection.

(8) Presence of any indwelling catheter or drainage tube (such as percutaneous nephrostomy tube, indwelling Foley catheter, bile drainage tube, or pleural/peritoneal/pericardial catheter); use of dedicated central venous access devices such as Port-A-Cath® or Hickman® catheters is allowed.

(9) Prior medication:

1. CD19-targeted therapy.
2. Use of chlorambucil or cladribine within 3 months prior to enrollment, or use of PEG-asparaginase within 3 weeks prior to enrollment.
3. Injection of live vaccines within 4 weeks prior to enrollment.
4. Donor lymphocyte infusion (DLI) within 28 days prior to enrollment.
5. Any drugs used for GVHD treatment within 4 weeks prior to enrollment (such as calcineurin inhibitors, methotrexate, mycophenolate, rapamycin, or salidroside), or use of immunosuppressive antibodies (such as anti-CD20, anti-tumor necrosis factor, anti-interleukin-6, or anti-interleukin-6 receptor) within 4 weeks prior to enrollment.
6. Immunostimulatory or immunosuppressive therapy within 4 weeks prior to enrollment (such as interferon-alpha, interferon-beta, IL-2, enoxaparin, efalizumab, alemtuzumab, tacrolimus, or mycophenolate).
7. Any systemic inhibitory/stimulatory immune checkpoint molecule therapy within 4 weeks prior to enrollment (e.g., ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc.).
8. Use of systemic cytotoxic drugs within 2 weeks prior to enrollment, including daily or weekly low-dose maintenance chemotherapy (such as cyclophosphamide, ifosfamide, bendamustine, chlorambucil, or mephalan, vincristine, etc.).
9. Long-acting growth factors within 14 days prior to single collection (such as pegfilgrastim) or short-acting growth factors within 5 days prior to single collection or drugs used for cell mobilization (such as G-CSF/PEG-CSF, plerixafor).
10. Receipt of radiotherapy within 2 weeks prior to enrollment.
11. Must avoid pharmacological doses of corticosteroids (>5 mg/day of prednisone or equivalent) and other immunosuppressive drugs within 7 days prior to single collection.
12. Use of venetoclax (BCL-2 inhibitor) within 4 days prior to single collection.
13. Short-acting targeted therapies (such as tyrosine kinase inhibitors) within 72 hours prior to single collection.
14. Use of idelalisib (oral PI3Kδ inhibitor) within 2 days prior to single collection.
15. Use of lenalidomide within 1 day prior to single collection.

(10) Active graft-versus-host disease (GVHD) using CIBMTR acute GVHD grading system ≥ grade 2 or requiring systemic steroids greater than physiological doses.

(11) History of autoimmune diseases in the past 2 years (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) resulting in end-organ damage or requiring systemic immunos uppressive/disease-modifying therapy.

(12) History of myocardial infarction, cardiac vascular surgery or stent implantation, unstable angina, or other clinically significant cardiac diseases within 12 months prior to enrollment.

(13) History of genetic syndromes associated with bone marrow failure, such as Fanconi anemia, Costello syndrome, Shwachman-Diamond syndrome, etc.

(14) Symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within the past 6 months. Subjects need to be on prophylactic anticoagulation.

(15) Past or present concurrent malignancies (excluding skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignancies that have not been treated and effectively controlled in the past five years).

(16) Use of other investigational medicinal products within 30 days prior to screening.

(17) Pregnant or lactating women of childbearing age, due to potential risks of chemotherapy to the fetus or infant. Women who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered of childbearing potential.

(18) Subjects unwilling to practice contraception from the agreement to treatment completion of conditional chemotherapy or CAR T infusion within 12 months (whichever is longer).

(19) Any medical conditions that may interfere with the safety or efficacy assessment of the study treatment.

(20) Subjects unlikely, in the investigator's judgment, to complete all protocol-required study visits or procedures, including follow-up, or comply with study requirements.

(21) Previous use of any CAR-T cell products or other genetically modified T cell therapies.

Ages: 18 Weeks to 70 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2039-12-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Up to 28 days from CAR-T infusion
  The proportion of patients receiving CAR-T cells who encounter dose-limiting toxicities (DLTs). Safety evaluations are performed in accordance with the NCI-CTCAE version 5.0 standards (Cytokine Release Syndrome and neurotoxicity will be graded based on ASTCT/ASBMT grading criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No